CLINICAL TRIAL: NCT07333222
Title: Prospective, Placebo-controlled Study on the Functional and Quality of Life Effects of the Mollii Neuromodulatory Suit in Patients With Stroke and Multiple Sclerosis
Brief Title: Functional and Quality of Life Effects of the Mollii Neuromodulatory Suit in Patients With Stroke and Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Somogy Megyei Kaposi Mór Teaching Hospital (Other)
Responsible Party: Principal Investigator, Tollár József, Head of Department, Somogy Megyei Kaposi Mór Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IG/4390-0/2025
Record Dates: First submitted 2025-12-19; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Multiple Sclerosis
Keywords: Stroke; Multiple Sclerosis; Mollii neuromodulation suit; Rehabilitation; Balance
MeSH Terms: conditions — Stroke; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mollii Group (Experimental): Receaving treatment with the stimulation program.
  Interventions: Other: the Mollii garment with active stimulation
- Control Group (Placebo Comparator): Receaving treatment without the stimulation program.
  Interventions: Other: Mollii neuromodulation garment, but the stimulation program is not activated (placebo)

INTERVENTIONS:
Other: the Mollii garment with active stimulation — Patients in the Intervention group attend therapy three days a week for four weeks, with each treatment lasting 60 minutes. In this group patients are fitted with the Mollii garment according to the same protocol, but in their case, active stimulation of the prescribed neuromodulation program is initiated.
  Arms: Mollii Group
Other: Mollii neuromodulation garment, but the stimulation program is not activated (placebo) — CG patients are fully equipped with the Mollii neuromodulation garment, but the stimulation program is not activated. The patient thus completes the therapy without the device's perceptible electrical stimulation, preserving the blinding effect of the placebo-controlled setup. The total treatment time, setup process, and therapeutic environment are the same as for the intervention group.
  Arms: Control Group

SUMMARY:
* Objective assessment of clinical symptoms resulting from stroke, as well as changes in mobility and quality of life, and determination of changes resulting from therapies
* Objective assessment of the quality of life, functionality, and clinical symptoms of patients with multiple sclerosis (MS) and determination of changes resulting from therapies
* Comparison of measured data from the two main neurological patient groups (stroke, multiple sclerosis) and follow-up of changes in relation to themselves and each other.
* Mapping the role of the placebo effect in neuromodulation devices by comparing subjective and objective outcomes.
* Analyzing the expectations and experiences of patients receiving placebo treatment using quality of life questionnaires.
* Analyzing the effects of the Mollii suit among subgroups of MS and stroke patients.
* Assessing the safety, possible side effects, and tolerability of the Mollii suit.
* Mapping changes in gait pattern due to the effects of therapy using 3D motion analysis.
* Examining the maintenance effects of neuromodulation during a 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* suffered a first ischemic stroke, diagnosed by a neurologist based on CT or MR imaging
* neurological examination revealed mobility and postural limitations
* confirmed multiple sclerosis diagnosed by a neurologist based on MRI imaging

Exclusion Criteria:

* multiple strokes in medical history
* systolic blood pressure less than 120 or higher than 160 mmHg
* orthostatic hypotension
* arotid artery stenosis
* severe heart disease
* hemophilia
* traumatic brain injury
* seizure disorder
* untreated diabetes
* abnormal electroencephalography
* abnormal blood panel
* use of sedatives
* irregular medication use
* severe aphasia (Western Aphasia Battery ≤ 25)
* severe visual or hearing impairment
* severe sensory dysfunction
* severe orthopedic problems
* other neurological conditions affecting motor function
* alcoholism
* drug use
* smoking after diagnosis of stroke
* unable to walk at least 10 m with or without assistance in 6 minutes
* BBS score ≤ 32
* BI score ≤ 70
* current participation in individual or group exercise program outside of standard physical therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | 4 weeks
  Functional autonomy, scaling 18-126 points. The lower the score, the less self-sufficient the patient is.
Barthel Index (BI) | 4 weeks
  Everyday activities, scaling 0-100 points. The higher the score, the better the self-sufficiency.

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) | 4 weeks
  Physical and psychological functions after stroke scaling 0-100 points, higher score means better post-stroke functions.
Multiple Sclerosis Impact Scale (MSIS-29) | 4 weeks
  Physical and psychological effects in MS, scaling 0-100 points, where higher scores mean greater disease impact.
Berg Balance Scale (BBS) | 4 weeks
  Measures balance, scaling 0-56 points, with lower scores suggesting good balance/indipandance.
Tinetti | 4 weeks
  Balance and walking, scaling 0-28 points, with lower scores indicating higher fall risk.
Timed Up and Go (TUG) | 4 weeks
  Measures functional mobility and fall risk, scaling 0-180 seconds. The less time, the lower the risk of falling.
6 minute walk test (6MWT) | 4 weeks
  Functional exercise capacity
10 meter walk test (10mWT) | 4 weeks
  Walking speed
Posturographic examination | 4 weeks
  Postural instability
3D motion analysis | 4 weeks
  Movement dynamics, gait

CONTACTS AND LOCATIONS:
Overall Officials: József Dr. habil Tollár, Principal Investigator — Somogy County Kaposi Mór Teaching Hospital
Locations (1):
- Somogy County Kaposi Mór Teaching Hospital, Kaposvár, Somogy County, Hungary

IPD SHARING:
Plan to Share IPD: No